CLINICAL TRIAL: NCT02166346
Title: Double-Blind, Placebo-Controlled Crossover Trial on the Safety and Efficacy of Sustained-Release Dalfampridine in Transverse Myelitis (Re-Launch)
Brief Title: Safety and Efficacy of Sustained Release Dalfampridine in Transverse Myelitis (Re-Launch)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00090799; NCT01446575 (obsolete NCT alias)
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Transverse Myelitis; Neuromyelitis Optica; Idiopathic Transverse Myelitis; Myelitis NOS
Keywords: Transverse myelitis
MeSH Terms: conditions — Myelitis, Transverse; Neuromyelitis Optica; Myelitis | interventions — 4-Aminopyridine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dalfampridine then Placebo (Experimental): All subjects were randomized for the first double-blinded 8-week part of the study to the dalfampridine group. Then subjects were crossed over to the placebo arm for another 8 weeks.
  Interventions: Drug: Dalfampridine; Drug: Placebo
- Placebo the Dalfampridine (Experimental): All subjects were randomized for the first double-blinded 8-week part of the study to the placebo arm. Then subjects were crossed over to the dalfampridine arm for another 8 weeks.
  Interventions: Drug: Dalfampridine; Drug: Placebo

INTERVENTIONS:
Drug: Dalfampridine — Dalfampridine 10 mg twice daily for 8 weeks
  Other Names: Ampyra
Drug: Placebo — Placebo pill 1 tablet twice daily for 8 weeks
  Other Names: Sugar pill

SUMMARY:
Transverse myelitis (TM) is an inflammatory disorder of the spinal cord that leads to disabilities of gait. Dalfampridine, a sustained-release potassium inhibitor has been shown to be effective in improving gait and other neurologic functions in multiple sclerosis. Dalfampridine has the potential to improve neurologic function in patients with transverse myelitis as this rare disorder shares a similar pathogenic process with multiple sclerosis. The in a clinical trial to test the efficacy of dalfampridine in TM.

The clinical trial that the investigators propose to conduct will focus on TM and will evaluate the dalfampridine in primary neurologic outcome, 25-foot timed walk, and several secondary outcomes including valid behavioral and neurophysiological tests.

This is a re-launch of the previous trial, which now includes additional behavioral and clinical testing.

DETAILED DESCRIPTION:
Fampridine (4-aminopyridine) is a potassium channel blocker that has been studied since the 1970s for its effect on amplifying conductivity in peripheral nerves, potentiating neurotransmitter release in muscles and increasing post-synaptic action potentials in the spinal cord. It was tested in other neurologic conditions over the next two decades and was found to have a limited therapeutic window due to the stimulation of seizures at high doses. The first randomized, placebo-controlled, double-blinded study of fampridine in 70 patients found significant improvements in a number of neurophysiological parameters while on fampridine compared to placebo. Since then, at least six additional studies on oral fampridine in Multiple Sclerosis (MS) were conducted and found to have some significant neurologic function. Although only a small incidence of seizure or altered mental status were reported in these studies, the concern about fampridine causing seizures remained a barrier in the acceptance of fampridine as an MS therapy in the general neurology community.

Recently, Biogen-Idec and Acorda have teamed up in the development of a sustained-release formulation of fampridine, dalfampridine, in which plasma concentrations of the drug and avoids toxic doses that lead to seizures. In two clinical trials, dalfampridine has been shown to be beneficial in two large cohorts of multiple sclerosis patients with noted improvements in gait and lower extremity muscle strength. Seizures were only seen in high doses of 20 mg or more whereas benefits were evident at the approved dose of 10 mg twice daily.

The Food and Drug Administration (FDA) approved dalfampridine for use in multiple sclerosis in 2009 based on the key study that evaluated gait by timed 25-foot walk. About 35-40% of study participants responded and this group improved their walking speed by about 20%.

The investigator's interest in dalfampridine is focused more narrowly on a subset of patients with a demyelinating disorder that is restricted to the spinal cord, transverse myelitis (TM), was not included in any previous human trials of dalfampridine. In contrast to MS, which affects the entire system, transverse myelitis affects the spinal cord and largely spares the brain. It is not associated with an increased risk of seizure.

Transverse myelitis is defined as an episode of inflammation in the spinal cord leading to disability at the level of the lesion and below. The majority of TM lesions strike the thoracic cord causing impairments in lower extremities. A single lesion is the cause of all of their symptoms. The goal of using dalfampridine in these patients is to amplify axonal conductance across the lesion. This would manifest as improved neurologic function involving the lower extremities including gait. This is a straightforward proof of concept model proving the mechanism of action of dalfampridine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of transverse myelitis confirmed by MRI
* Gait impairment defined as a baseline timed 25-foot walk of at least 5 seconds and no more than 60 seconds.
* Age 18-70.

Exclusion Criteria:

* Diagnosis of any of the following concurrent conditions: spinal dural arteriovenous malformation, multiple sclerosis, infectious myelitis and recurrent transverse myelitis of any etiology. Subjects with a positive NMO-Immunoglobulin G (IgG) biomarker test will be permitted to join the study as long as the there is only a history of monophasic, and not recurrent, TM.
* History of seizure(s).
* Pregnancy or positive pregnancy test (mandatory test for all women aged 18-55 to be done at first screening visit).
* Known use or allergy to dalfampridine or any other formulation of 4-aminopyridine.
* Patients unable to walk.
* Patients with history of severe alcohol or drug abuse, severe psychiatric illness such as severe depression, poor motivational capacity, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as equivalent to a mini-mental state exam score of 23 or less).
* Patients with severe uncontrolled medical problems (e.g. hypertension, cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, claudication, uncontrolled epilepsy or others).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2017-01-08 (Actual); Study Completion 2017-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levy, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dalfampridine Then Placebo: All subjects were randomized for the first double-blinded 8-week part of the study to the dalfampridine group. Then subjects were crossed over to the placebo arm for another 8 weeks.
  Dalfampridine: Dalfampridine 10 mg twice daily for 8 weeks Placebo: Placebo pill 1 tablet twice daily for 8 weeks
- Placebo Then Dalfampridine: All subjects were randomized for the first double-blinded 8-week part of the study to the placebo arm. Then subjects were crossed over to the dalfampridine arm for another 8 weeks.
  Placebo: Placebo pill 1 tablet twice daily for 8 weeks Dalfampridine: Dalfampridine 10 mg twice daily for 8 weeks
Period: Screening and Randomization
Arm/Group | Dalfampridine Then Placebo | Placebo Then Dalfampridine
Started | 12 | 12
Completed | 8 | 8
Not Completed | 4 | 4
Period: Intervention - Phase 1
Arm/Group | Dalfampridine Then Placebo | Placebo Then Dalfampridine
Started | 8 | 8
Completed | 8 | 6
Not Completed | 0 | 2
Period: Intervention - Phase 2 (After Crossover)
Arm/Group | Dalfampridine Then Placebo | Placebo Then Dalfampridine
Started | 8 | 6
Completed | 7 | 6
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: 24 participants consented, 8 were excluded = 16 enrolled. Of the 16 enrollees, 3 withdrew = 13 completers.
Groups:
- Whole Study Population: This is a crossover trial. At baseline prior to randomization into an intervention, the baseline measures are provided.
Arm/Group | Whole Study Population
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 55 [33 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Duration of Disease [Mean (Full Range); unit: years] | 7.2 [3 to 31]
Expanded Disability Status Scale score [Mean (Full Range); unit: units on a scale] — In this scale, 0 is normal and 10 is dead. Additional information can be found here: https://www.mstrust.org.uk/a-z/expanded-disability-status-scale-edss
  units on a scale | 4.9 [3.5 to 6]
Lesion location within spinal cord [Count of Participants; unit: Participants]
  Cervical | 4
  Cervicothoracic | 5
  Thoracic | 4
Lesion length by MRI [Mean (Full Range); unit: vertebral lengths] — Vertebral length is defined as the number of vertebrae between the top of the T2 hyper intense lesion by MRI and the bottom of the lesion visualized on the middle sagittal section.
  vertebral lengths | 6 [2 to 13]

OUTCOME MEASURES:

1. Primary Outcome: Walking Speed During Timed 25-foot Walk
Description: In this cross-over study, walking speed was recorded 4 times for each subject while in both the dalfampridine and placebo arms. The results average all of the times while on damfampridine and compares them to the average of the times while on placebo.
Time Frame: Every 2 weeks during each 8 week intervention
Population: In this cross-over study, walking speed was recorded 4 times for each subject while in both the dalfampridine and placebo arms. The results average all of the times while on damfampridine and compares them to the average of the times while on placebo.
Measure: Mean (Full Range); unit: feet/second
Groups:
- Dalfampridine: All subjects will be randomized for the first double-blinded 8-week part of the study with 25-foot timed walking assessments every 2 weeks. Then subjects will be crossed over to the other therapy (drug or placebo) for another 8 weeks.
  Dalfampridine: Dalfampridine 10 mg twice daily for 8 weeks
- Placebo: Placebo controlled arm.
  Placebo: Placebo pill 1 tablet twice daily for 8 weeks
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 13 | 13
feet/second
  Change from baseline to 2 weeks | 0.3342 [0.0975 to 0.5709] | 0.4745 [0.2294 to 0.7195]
  Change from baseline to 4 weeks | 0.4593 [0.2071 to 0.7114] | 0.1743 [-0.06251 to 0.4111]
  Change from baseline to 6 weeks | 0.5445 [0.1018 to 0.9872] | 0.5697 [0.1596 to 0.9799]
  Change from baseline to 8 weeks | 0.3803 [-0.0113 to 0.7719] | 0.2101 [-0.1757 to 0.5959]

2. Secondary Outcome: Upper and Lower Extremity Muscle Strength Measurements
Description: Upper and lower extremity muscle strength measurements, using a hand held dynamometer, at the beginning and end of each arm. Change in muscle strength between baseline and end (8 weeks) of each intervention are provided.
Time Frame: baseline and end (8 weeks) of each intervention
Measure: Mean (95% Confidence Interval); unit: Pounds
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 13 | 13
Pounds
  Supine Left Hip Flexor | .6420 [-7.3278 to 8.6118] | -0.05187 [-6.3646 to 6.2609]
  Supine Right Hip Flexor | 2.5774 [-2.4644 to 7.6192] | 2.854 [-1.31 to 7.018]
  Prone Left Hip Flexor | 3.286 [-6.5985 to 13.1717] | -1.497 [-10.053 to 7.0572]
  Prone Right Hip Flexor | 3.9752 [-6.8518 to 14.8022] | -4.4162 [-13.7929 to 4.9604]
  Left Grip | 3.1594 [-4.844 to 11.1628] | -2.9007 [-10.7863 to 4.9849]
  Right Grip | -1.3602 [-6.7146 to 3.9942] | 2.1665 [-3.1048 to 7.4378]

ADVERSE EVENTS:
Arm/Group | Dalfampridine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 4/13 | 5/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalfampridine (N=13) | Placebo (N=13)
Urinary urgency (Renal and urinary disorders) | 4 (4) | 5 (5)
Insomnia (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Weakness (Nervous system disorders) | 4 (4) | 2 (2)
Fatigue (Nervous system disorders) | 4 (4) | 4 (4)
Muscle stiffness (Nervous system disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No